CLINICAL TRIAL: NCT00424567
Title: TRC Autologous Bone Marrow Cells for the Treatment of Appendicular Skeletal Fracture Non-Union
Brief Title: Feasibility Study of Aastrom Tissue Repair Cells to Treat Non-Union Fractures.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed early for business reasons (not safety reasons)
Sponsor: Vericel Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI 55-0503-1
Expanded Access: Available
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Fracture, Ununited; Pseudarthrosis
Keywords: Fracture; non union fracture; ununited fracture; pseudarthrosis
MeSH Terms: conditions — Fractures, Ununited; Pseudarthrosis; Fractures, Bone

INTERVENTIONS:
Procedure: Fracture surgery
Drug: Cultured Bone Marrow Tissue

SUMMARY:
The purpose of this multi-center study is to obtain clinical data to substantiate that Aastrom TRC autologous bone marrow cells will regenerate bone in patients with established (appendicular skeletal) non union fractures, when used with one of the commonly employed commercially available allograft chip matrices.

DETAILED DESCRIPTION:
The current standard of care for regeneration of atrophic long bone fracture non-union is autologous bone and marrow chiseled from the patient's iliac crest in open surgery under general anesthesia. This method for harvesting bone and marrow is associated with substantial morbidity of long-term pain, the possibility of deep-seated infection at the site of the bone harvest and other indirect consequences such as extended time of surgery, substantial expense and the potential for blood transfusion. The procedure is also associated with a bone graft failure rate of at least 20%.

Due to the substantial morbidity resulting from the aggressive open surgical procedure, alternatives are sought. Current alternatives to autologous bone include commercially available synthetic, xenograft and allograft matrices, either used alone or combined with bone autograft. Cell-free substitutes, such as matrices combined with platelet rich plasma or recombinant bone morphogenic proteins for osteoinductivity, are also used. These alternatives, although less morbid than a full bone harvest, have not yet been stringently determined to be equivalent. Therefore, there is a continuing search for additional improved alternatives.

Aastrom Biosciences, Inc. has developed a unique process for growing human bone marrow, including the early stem cell populations, from small samples of percutaneously aspirated bone marrow. The process is carried out in the AastromReplicell Cell Production System (ARS).

The study will be performed to obtain clinical data to substantiate that Aastrom TRC autologous bone marrow cells will regenerate bone in patients with established non union fractures, when used with one of the commonly employed commercially available allograft chip matrices.

The bone marrow cells will be obtained by a brief, percutaneous, small volume aspiration (approximately 30 - 50 ml) from the posterior iliac crest obtained under local and conscious sedation. Percutaneous marrow aspiration is substantially less morbid and time consuming than the current open surgical process of bone autograft harvest.

The study will treat up to 36 patients (11 in the first group and 25 in a second group).

Patients will be treated using standard surgical procedures for the treatment of non union fractures (including commonly used hardware needed to stabilize the fracture). The processed cells will be mixed with commercially available bone matrix during surgery and placed in the area of the fracture.

Patients will be monitored for 12 months following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Type IIIA or IIIB fracture
* Fracture gap < 6 cm.
* Distance of > 4 cm from joint
* No clinical signs of infection at the wound site or fracture site.
* Adult patients >18 years of age.
* Male patients or female patients who are not pregnant or lactating.
* Patients must have normal organ and marrow function as defined below:

  1. Leukocytes >=3000/microliters
  2. Absolute neutrophil count >=1500/microliters
  3. Platelets >=100,000/microliters
  4. AST (SGOT)/ALT (SGPT) <2.5 x institutional limits
  5. Creatinine within normal limits or creatinine clearance calculated)>=60 mL/min/1.73 square miter with creatinine above institutional normal.
* Patients able to give informed consent

Exclusion Criteria:

* Other long bone fractures, e.g clavicle
* Patients unable to discontinue ethanol use after surgery including those requiring pharmacologic adjuvant assistance.

  1. Although not an exclusion criteria, the attending physician shall discuss with the patient the advantages of discontinuing smoking cigarettes and/or cigars during the term of the study including discontinuing the use of pharmacologic adjuvant assistance such as nicotine suppression.
  2. The use or discontinuance of ethanol and/or cigarettes/cigars will be noted in the patient's case report forms.
* Patients who require corticosteroid anti-inflammatory therapy after surgery.
* Patients with genetic metabolic bone disease such as hypophosphatasia, or metabolic bone disorders such as primary or secondary hyperparathyroidism caused by chronic renal insufficiency or other disorders.
* Patients unable to tolerate general anesthesia defined as an ASA criteria of 0 or 1.
* Patients on systemic antibiotics for suspected wound or fracture site infection.
* Patients with diabetes.
* Glasgow score of < 13.
* Injury severity score of > 25.
* Allergy to protein products derived from mammalian sources (horse, bovine or porcine) required in the ex-vivo cell production process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-10; Study Completion 2007-06

PRIMARY OUTCOMES:
The primary endpoint will be the proportion of patients with demonstrated healing, including bone formation, at 12 months (or until completely healed) from surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Jimenez, MD, Principal Investigator — Illinosis Bone and Joint Institute; James Goulet, MD, Principal Investigator — University of Michigan; Thomas Lyon, MD, Principal Investigator — Lutheran Medical Center; Nowinski, MD, Principal Investigator — Corewell Health East
Locations (4):
- United States (4):
  - Illinois Bone and Joint Institute, Des Plaines, Illinois
  - University of Michigan Medical School, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Lutheran Medical Center, Brooklyn, New York